CLINICAL TRIAL: NCT04071626
Title: The EMMED-HF Study: Evaluating Metabolic Mechanisms of Ertugliflozin in Diabetes & Heart Failure
Brief Title: Evaluating Metabolic Mechanisms of Ertugliflozin in Diabetes & Heart Failure
Acronym: EMMED-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Trevor Jenkins, Assistant Professor of Medicine, Department of Medicine, Case Western Reserve University / UH Cleveland Medical Center, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20190016
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure, Diastolic; Diabetes Mellitus, Type 2
Keywords: ertugliflozin; SGLT2 inhibtion; Cardiovascular Diseases; Sodium-Glucose Transporter 2 Inhibitors; Glucose Metabolism Disorders; Physiological Effects of Drugs; Diabetes Mellitus; Diabetes Mellitus, Type 2; Endocrine System Diseases
MeSH Terms: conditions — Heart Failure, Diastolic; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Glucose Metabolism Disorders; Diabetes Mellitus; Endocrine System Diseases | interventions — ertugliflozin

STUDY DESIGN:
Intervention Model Description: Parallel assignment, active controlled, single center experimental design.
Who Masked: Participant, Care Provider
Masking Description: Single-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ertugliflozin Treatment Arm (Experimental): Ertugliflozin 5 mg tablet once a day for 12 weeks
  Interventions: Drug: Ertugliflozin 5 mg
- Placebo (Placebo Comparator): Placebo tablet once a day for 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin 5 mg once a day for 12 weeks
  Arms: Ertugliflozin Treatment Arm
Drug: Placebo oral tablet — Placebo oral tablet once a day for 12 weeks
  Arms: Placebo

SUMMARY:
This clinical trial will determine if subjects with heart failure with preserved ejection fraction (HFpEF) and type 2 diabetes mellitus (DM2) receiving sodium-glucose cotransporter 2 (SGLTi2) inhibitor therapy (ertugliflozin) alters cardiac metabolism compared to placebo in a single blinded (to subject), randomized, parallel group, active controlled, single center experimental design.

DETAILED DESCRIPTION:
The results of recent sodium-glucose cotransporter 2 (SGLT2) inhibitor therapy clinical trials demonstrate clinically significant reductions in cardiovascular endpoints (myocardial infarction, cardiac death, heart failure hospitalization). SGLT2 inhibition appears to exert cardiovascular protection through pleiotrophic effects involving both the myocardium and peripheral organs but the primary pathway of risk reduction of heart failure incidents has not been elucidated. SGLT2 inhibitors induce a loss of 50-100 grams of glucose through urinary excretion daily. There is a compensatory increase in ketone body production in the liver after initiation of SGLT inhibition. Ketone bodies are the most energy efficient myocardial fuel source and reduce myocardial oxidative stress when consumed as the primary energy substrate. Inducing a shift to ketone body metabolism to improves cardiac diastolic performance suggests a unifying paradigm of direct myocardial effect and peripheral metabolic flexibility through which SGLT2 inhibition mediates myocardial protection in HFpEF.

Specific Aims Aim 1: Determine if 12 weeks of SGLTi2 therapy improves peak exercise oxygen uptake compared to placebo. We will perform cardiac MRI exercise testing (CPET-ExMR) before and & post 12 weeks of therapy to measure cardiopulmonary fitness by metabolic cart gas exchange and left ventricular myocardial mass.

Aim 2: Evaluate the short term (12 weeks effect of SGLTi on metabolic flexibility in HFpEF compared to baseline function and control group. We will measure glucose and lipid metabolism response to SGLT2 inhibition. Serum samples of glucose and ketone bodies (β-hydroxybutyrate) will be assessed before & post 12 weeks of therapy. Serial serum samples will allow us to generate metabolomics profiles before and after treatment. This experimental design will provide insight into ketone body production, peripheral glucose flux, and circulating lipoparticles in response to SGLTi therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old but < 75 years old
* No HF hospitalization within 6 months
* Overweight or Obesity defined as BMI > 29 but < 42
* History of insulin resistance or T2DM and on oral diabetes agents other than SGLT2i (HgbA1c > 5.8% and < 10.5%)
* EF calculated based on a recent echo/cath/nuclear study at screening (pre-enrollment) > 50%
* Stable HFpEF (HF with preserved ejection fraction) medications use of 3 months with no plans to changes or add medications for at least 12 weeks course of the study)

Exclusion Criteria:

* Acute HFpEF hospitalization within 6 months of enrollment.
* CKD stage 4 or 5 (eGFR < 30 ml/min by CKD-EPI equation).
* Other known causes of HF including poorly controlled hypertension (SBP >160 mm Hg) or ischemic cardiomyopathy (etc).
* Anemia (Hgb < 11.0 mg/dL for women and < 12.0 mg/dL for men) or severe thrombocytopenia (platelets < 50,000 mm3)
* Anticipated changing of HF medication during anticipated study period.
* HFREF (LV EF < 50%).
* Acute coronary syndrome, transient ischemic attack, CVA or critical limb ischemia during the last 6 months or coronary/peripheral revascularization within the last 3 months. Severe life threatening illness or live expectancy < 6 months.
* Contraindications to MRI (metallic implants, severe claustrophobia) or treadmill exercise (limb amputation, severe osteoarthritis or equivalent functional mechanical limitation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor L Jenkins, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertugliflozin Treatment Arm | Placebo
Started | 5 | 4
Completed | 4 | 2
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin Treatment Arm | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2, ml/kg/Min, as Measured by Metabolic Gas Exchange
Description: The difference in peak oxygen uptake as measured by peak VO2 (ml/kg/min) between ertugliflozin and placebo as measured at baseline and after 12 weeks of treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Peak VO2, ml/kg/min
Arm/Group | Ertugliflozin Treatment Arm | Placebo
Number analyzed (Participants) | 4 | 2
Peak VO2, ml/kg/min | -0.6 (1.13) | -0.1 (1.23)

2. Secondary Outcome: Left Ventricular Mass Index (gm/m2), as Measured by Cardiac MRI
Description: The difference in LV mass index (gm/m2) measured by cardiac MRI between ertugliflozin and placebo as measured at baseline and after 12 weeks of treatment
Time Frame: 12 weeks
Population: Data not collected.
Arm/Group | Ertugliflozin Treatment Arm | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Serum Ketone Bodies (Betahydroxybutyrate)
Description: The difference in serum ketone bodies (betahydroxybutyrate) levels between ertugliflozin and placebo as measured at baseline and after 12 weeks of treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ertugliflozin Treatment Arm | Placebo
Number analyzed (Participants) | 4 | 2
mmol/L | -0.045 (0.078) | -0.018 (0.028)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ertugliflozin Treatment Arm | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT04071626/Prot_SAP_000.pdf